CLINICAL TRIAL: NCT01227109
Title: Procalcitonin as a Marker of Infection in Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Herlev Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Anders Mellemgaard, Herlev University Hospital
Other Study IDs: Procalcitonin-one
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Infections; Cancer; Procalcitonin; C Reactive Protein
Keywords: Infections; Cancer; Procalcitonin; C reactive protein
MeSH Terms: conditions — Infections; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be drawn for CRP and procalcitonin analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With infection: This group consist of cancer patients with a bacterial infection
- Without infection: This is a group of cancer patients without infection

SUMMARY:
Infections pose a serious threat to cancer patients in chemotherapy. Prompt diagnosis and treatment is of paramount importance as infections may be life-threatening in immune-compromised individuals. Traditionally, the C-reactive protein (CRP) has been used as a marker of infection. However, the CRP is also often elevated in cancer patients and as a marker CRP may be unreliable in cancer patients. Other markers for infection includes procalcitonin which has been showed to be of some value for the diagnose of bacterial infections.

This study examines procalcitonin as a potential marker of bacterial infection in cancer patients.

DETAILED DESCRIPTION:
Purpose of the study:

Is pro calcitonin a marker for bacterial infection in cancer patients? Is pro calcitonin better than C-reactive-protein to identify cancer patients with a bacterial infection?

Background:

Infections, in particular bacterial, pose a major threat to cancer patients as treatment related immuno-suppression and general weakness increase risk and severity of infections. Prompt identification of patients with a bacterial infection is necessary. Traditionally, fever, leucocytosis and elevated c-reactive protein (CRP) have been used in the evaluation in patients with suspected infection. How-ever, fever may be reduced by analgesics and steroids, leucocytes may be decreased due to anticancer therapy and CRP is in some cases elevated by the cancer disease as such. The diagnosis of bacterial infection is thus more difficult in cancer patients. Recently, pro-calcitonin (PCT) (her dækker maja's godt)

Design of the study:

Two groups will be included in this study:

Group I includes patients in anti-cancer therapy including chemo and radiotherapy, targeted treatment and radiotherapy but not hormone treatment, and without any sign of infection defined as temperature < 38 C and no focal symptoms of infections. Vital signs are noted and blood tests for haematology, CPR and PCT are drawn. Details about cancer type, stage, treatment history of infections less than 1 month prior and co-morbidity are registered. Data from this cohort will be used to assess median CRP and PCT among non-infected cancer patients. Forty patients will be included.

Group II includes patients in anti-cancer therapy including chemo and radiotherapy, targeted treatment and radiotherapy but not hormone treatment, who is hospitalized with suspected infection (temp> 38 last 24 hours). At the time of hospitalization, vital signs are noted and blood tests for haematology, CPR and PCT are drawn. Details about cancer type, stage, treatment history of infections less than 1 month prior and co-morbidity are registered. All hospitals records are reviewed after discharge to determine if a certain diagnosis of infection (positive bacteriology), probable infection (negative bacteriology but clinical course consistent with bacterial infection) or non infection was made. Data from this cohort will be used to assess the role of CRP and PCT in prediction of bacterial infection. Forty patients will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

Gr I: In-patients in anticancer therapy for a solid cancer with confirmed bacterial infection Gr II: Patients in anticancer therapy without any signs or symptoms of infection.

Both groups: Informed consent

Exclusion Criteria:

None

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Two groups of 40 patiens each, one with bacterial infection, the other without any signs or symptoms of infection
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of procalcitonin elevation in cancer patients with or with out infection | less than 60 days
  The mean procalcitonin value will be compared between two groups of cancer patients with and with-out infections respectively.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Herlev University Hospital, Copenhagen
  - Herlev hospital, Herlev

REFERENCES:
- [Derived] Diness LV, Maraldo MV, Mortensen CE, Mellemgaard A, Larsen FO. Procalcitonin and C-reactive protein as markers of bacterial infection in patients with solid tumours. Dan Med J. 2014 Dec;61(12):A4984. PMID 25441735